CLINICAL TRIAL: NCT03864107
Title: Investigating the Possible Link Between Habitual Diet, Physical Activity, Sleeping Patterns, Obesity Status and Age With Gut Bacterial Composition, Gut Barrier Function, Metabolic Endotoxemia, Systemic Inflammation and Glycaemic Control.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Carl Hulston, Senior Lecturer Nutrition and Metabolism, Loughborough University
Other Study IDs: R18-P206
Record Dates: First submitted 2019-02-14; First posted 2019-03-06 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Metabolic Syndrome; Insulin Resistance
Keywords: Glycaemic Control; Gut Permeability; Gut Microbiota; Metabolic Endotoxemia; Metabolic Health
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood plasma/ serum, urine, faeces, peripheral blood mononuclear cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the UK, 25% of the adults are affected by metabolic syndrome (NHS, 2016). Metabolic syndrome is a cluster of different conditions including: hyperglycaemia, insulin resistance hypertriglyceridemia, dyslipidaemia and hypertension. Such individuals also have increased risk of developing type 2 diabetes and cardiovascular disease. The factors contributing to the development of metabolic syndrome are potentially numerous and understudied in humans, with much of what we think we know coming from animal research. Recent animal studies have pointed towards gut health playing a role in metabolic health. More specifically it has been suggested that changes in the composition of the gut microbiota may drive insulin resistance and type 2 diabetes through a mechanism that is linked to increased gut permeability and the development of metabolic endotoxemia and inflammation. Yet, this link has not been confirmed in humans. This research will look at the relationship between diet, physical activity, sleeping patterns, obesity status and age etc. and measures of gut bacterial composition, gut barrier function and metabolic health. Findings will provide us with new insights on the effect of different physiological and behavioural/ lifestyle variables on gut health and metabolic function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-70 years
* BMI 18.5-50 kg/m2
* Not taking antibiotics and antimicrobial drugs for at least three months
* Both physically active and sedentary individuals will be eligible to take part in the study
* Weight stable (±5kg) for at least 6 months

Excusion Criteria:

* No cardiometabolic (e.g. heart disease, high blood pressure) or inflammatory illness
* Smokers (including the use of vaporisers and e-cigarettes)
* Taking anti-inflammatory drugs (excluding aspirin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women living in and around Loughborough, Leicestershire, United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control / Whole body insulin sensitivity index | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed by oral glucose tolerance test
Systemic Markers of Metabolic Endotoxemia (for example LBP determined using an ELISA) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples

SECONDARY OUTCOMES:
Gut permeability | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Urine samples will be used to assess the ratio of lactulose to mannitol excretion
Anthropometric Measurements (for example height and weight that will be aggregated to report BMI in kg/m^2) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Measured using standard equipment
Fasting Serum Lipid Profile (for example total, HDL and LDL cholesterol, TAG, free fatty acids measured by spectrophotometric assay) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples
Systemic Markers of Inflammation (for example IL-6, CRP determined using an ELISA/ spectrophotometric assay) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples
Systemic Markers of Oxidative Stress (for example protein carbonyls, glutathione and redox enzymes by ELISA/ spectrophotometric assay (in sub-cohort of participants not taking high-dose antioxidant supplements) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples
Fasting hormone concentration (for example ghrelin, leptin measured by ELISA) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples
Characterisation of immune cell migratory capacity using an ex vivo model (in a sub-cohort of obese participants only) | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples by flow cytometry analysis
Characterisation of immune cell populations (monocyte subsets) from peripheral blood mononuclear cells | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed following the collection of fasted blood samples by flow cytometry analysis
Dietary intake | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Assessed via a Food Frequency Questionnaire (FFQ)
Fasting blood pressure | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Systolic and diastolic blood pressure and central blood pressure, measured in triplicate using a Mobil-O-Graph following 20 min period of seated rest
Fasting arterial stiffness | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Pulse wave analysis and velocity, measured in triplicate using a Mobil-O-Graph following 20 min period of seated rest
Step count | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Habitual daily step count as measured by pedometer for 7 consecutive days prior to the first experimental session
Self-reported activity | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Participants will complete the International Physical Activity Questionnaire to measure participants' time spent in physical activity.
Sleeping pattern | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Habitual sleep pattern will be assessed by sleep diary 7 consecutive days prior to the first experimental session
Functional tests | Cross-sectional (all outcome measures will be collected within a 4 week period)
  To be assessed by handgrip strength (measured in force) and timed sit-to-stand movements (measured as time in seconds to perform 5 sit-to-stand movements followed by the maximum number of movements that can be completed in 60 seconds)
Questionnaires | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Morningness and Eveningness questionnaire; Mood state
Urinary metabolomics | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Urine samples will be used for metabolic profiling of excreted metabolites
Microbiome analysis | Cross-sectional (all outcome measures will be collected within a 4 week period)
  Faecal samples will be used to analyse gut microbiota composition through the 16S ribosomal RNA gene sequencing technique

CONTACTS AND LOCATIONS:
Overall Officials: Carl Hulston, PhD, Principal Investigator — Loughborough University
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough, Leicestershire, United Kingdom